CLINICAL TRIAL: NCT04232527
Title: Prospective Cohort Study, Follow-up of Subjects Over Long Periods, Assessment of Test Reliability in Predicting Injury Risk
Brief Title: Dynamic Balance, Flexibility and Agility as Predictors of Lower-extremity Injury in Football Players
Status: Completed | Type: Observational
Sponsor: Dragan Mijatović (Other)
Responsible Party: Sponsor-Investigator, Dragan Mijatović, Master of Physiotherapy, Postgraduate Study in Health Sciences, University of Mostar
Organization: University of Mostar (Other)
Other Study IDs: DMijatovic
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: LOWER-LIMB INJURY
Keywords: Dynamic balance; Stretching; Flexibility; Agility
MeSH Terms: conditions — Leg Injuries | interventions — Sitting Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Professional Footballers: About 110 players (out of about 400 competing in the Premier League of Bosnia and Herzegovina) would be included in the research.
  Interventions: Diagnostic Test: Y Balance Test; Diagnostic Test: Sit and Reach Test; Diagnostic Test: "Maximum Legs Abduction" Test; Diagnostic Test: S_RAG (reactive agility)" Test; Diagnostic Test: S_CODS (change of direction speed) Test

INTERVENTIONS:
Diagnostic Test: Y Balance Test — The footballer will place one foot on the stationary platform of the test set during the test so that the top of the sneaker does not exceed the starting line. The second foot, or the tip of the foot, will push the movable part of the platform down the measuring tube, which is marked by half-inch intervals. Any lifting of the standing leg on the heel, on the toes or loss of balance will be considered a mistake and the attempt will be repeated. Mobility will be tested through 3 trial and 3 valid measurements of the lower limbs in the anterior, posteromedial, and posterolateral directions. The arms should rest on the hips.
Diagnostic Test: Sit and Reach Test — This test involves sitting on the floor with your legs stretched straight forward. Shoes should be removed. The feet themselves are set straight against the box. Both knees must be stretched. With the palms facing down and the palms side-by-side or side-by-side, the subject approaches the measurement line as far as possible. It is important to keep your hands in the same position level, not that one reaches further than the other. Once the subject has reached the maximum distance, hold this position for one to two seconds and record the distance.
Diagnostic Test: "Maximum Legs Abduction" Test — Seated legs abduction is a test to assess the flexibility of the groin region. Respondent without the shoe sits with its back and head resting against the wall. As a sign, the subject extends the legs (stretches) to the maximum extent. During the test, the legs should not be bent at the knee joint.
Diagnostic Test: S_RAG (reactive agility)" Test — The test consist of fast-moving forward, and a change of direction conditioned by visual stimuli.
Diagnostic Test: S_CODS (change of direction speed) Test — S_CODS (change of direction speed) is a test that allows athletes to outperform their opponents in situations where they can pre-define a movement pattern.

SUMMARY:
This research investigates the reliability of tests to assess injury risk. Participants will be tested at the beginning of the survey and will be monitored for over 5 months. Participants will take 4 types of tests related to dynamic balance, flexibility, and agility. Subsequently, the relationship between test results and the incidence of injury in the subjects will be analyzed. If the tests prove reliable, they will be included in standard tests to assess the risk of injury to football players.

DETAILED DESCRIPTION:
Too often, injuring athlete results in a large amount of money being spent on rehabilitation. In a world of sports where the speed of recovery means a lot, ways are sought first and foremost to minimize the frequency of non-contact injuries. To prevent certain things, it is important to know the initial state, therefore, to see if certain factors at the outset indicate to us that there is a certain imbalance that can result in the injury. Since we live in a country where sports clubs are unable to spend large amounts of money on rehabilitation, it would be of great benefit to find reliable tests that can help to prevent an injury. Studies have shown that tests of balance, flexibility, and agility can help to prevent injury to football players in other countries. The same tests will be applied to Premier League footballers in Bosnia and Herzegovina and their effectiveness in assessing the degree of risk of lower limb injuries will be tested. If they prove reliable, they can become a standard in the prevention of these injuries, that is, they will help in the development of injury prevention programs, which would be of great benefit to both clubs and football players.

The study aims to determine whether dynamic balance and flexibility tests can be used as reliable predictors of lower limb injuries in football players and whether reduced agility influences the increased risk of injury.

ELIGIBILITY:
Inclusion Criteria:

* Professional players
* Age above 18 years
* Voluntary access to research

Exclusion Criteria:

* Age under 18,
* Refusal to take the research,
* Remaining in the club until the end of the examination,
* Errors in keeping records of injuries by responsible persons,
* Injuries to the lower limbs in the last ten days,
* Vestibular disorders.

Ages: 18 Years to 40 Years | Sex: Male
Age Groups: Adult
Study Population: About 110 players (out of about 400 competing in the Premier League of Bosnia and Herzegovina) would be included in the research.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-08-26 (Actual)

PRIMARY OUTCOMES:
The incidence | 5 month
  The main outcome measure is the incidence, that is, the number of newly injured players over almost five months.

SECONDARY OUTCOMES:
Questionnaire to evaluate the current situation with lower limb injuries in football players | 5 minutes
  It consists of 20 questions that ask about the condition of the lower limbs in tested football players.
Y balance test | 15 minutes
  Mobility will be tested through 3 trial and 3 valid measurements of the lower limbs in the anterior, posteromedial, and posterolateral directions.
Sit and Reach test | 5 minutes
  The Sit and Reach Test is a common muscle and lower back flexion test and is now widely used as a general flexibility test.
Maximum legs abduction Test | 5 minutes
  A seat abduction test is a test to assess the flexibility of the groin regions. The footballer extends his legs as far as possible (stretches). The distance between the inner malleolus is measured in centimeters tape.
S_RAG (reactive agility) Test | 10 minutes
  S_RAG (reactive agility) Test is emphasized when athletes perform a change of direction while responding to an external visual stimulus.
Measuring the length of the legs | 2 minutes
  Anthropological measures will be taken (from the spin of the iliac anterior superior to the middle of the inner malleolus).
S_CODS (change of direction speed) Test | 2 minutes
  S_CODS (change of direction speed) is a test that allows athletes to outperform their opponents in situations where they can pre-define a movement pattern.

CONTACTS AND LOCATIONS:
Overall Officials: Damir Sekulić, PhD, Study Chair — KIF Split
Locations (1):
- NK "Široki Brijeg", Široki Brijeg, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones BH, Cowan DN, Tomlinson JP, Robinson JR, Polly DW, Frykman PN. Epidemiology of injuries associated with physical training among young men in the army. Med Sci Sports Exerc. 1993 Feb;25(2):197-203. PMID 8450721
- [Background] van Mechelen W. Running injuries. A review of the epidemiological literature. Sports Med. 1992 Nov;14(5):320-35. doi: 10.2165/00007256-199214050-00004. PMID 1439399
- [Background] Kinzey SJ, Armstrong CW. The reliability of the star-excursion test in assessing dynamic balance. J Orthop Sports Phys Ther. 1998 May;27(5):356-60. doi: 10.2519/jospt.1998.27.5.356. PMID 9580895
- [Background] Greenberg ET, Barle M, Glassmann E, Jung MK. INTERRATER AND TEST-RETEST RELIABILITY OF THE Y BALANCE TEST IN HEALTHY, EARLY ADOLESCENT FEMALE ATHLETES. Int J Sports Phys Ther. 2019 Apr;14(2):204-213. PMID 30997273
- [Background] Lee SK, Ahn SH. Effects of balance evaluation comparison of dynamic balance and Y balance. J Exerc Rehabil. 2018 Dec 27;14(6):939-943. doi: 10.12965/jer.1836494.247. eCollection 2018 Dec. PMID 30656152
- [Background] Sheppard JM, Young WB. Agility literature review: classifications, training and testing. J Sports Sci. 2006 Sep;24(9):919-32. doi: 10.1080/02640410500457109. PMID 16882626
- [Background] Sekulic D, Spasic M, Mirkov D, Cavar M, Sattler T. Gender-specific influences of balance, speed, and power on agility performance. J Strength Cond Res. 2013 Mar;27(3):802-11. doi: 10.1519/JSC.0b013e31825c2cb0. PMID 22580982
- [Background] Brunner R, Friesenbichler B, Casartelli NC, Bizzini M, Maffiuletti NA, Niedermann K. Effectiveness of multicomponent lower extremity injury prevention programmes in team-sport athletes: an umbrella review. Br J Sports Med. 2019 Mar;53(5):282-288. doi: 10.1136/bjsports-2017-098944. Epub 2018 Sep 10. PMID 30201793
- [Background] Robinson RH, Gribble PA. Support for a reduction in the number of trials needed for the star excursion balance test. Arch Phys Med Rehabil. 2008 Feb;89(2):364-70. doi: 10.1016/j.apmr.2007.08.139. PMID 18226664
- [Background] Sisic N, Jelicic M, Pehar M, Spasic M, Sekulic D. Agility performance in high-level junior basketball players: the predictive value of anthropometrics and power qualities. J Sports Med Phys Fitness. 2016 Jul-Aug;56(7-8):884-93. Epub 2015 May 5. PMID 25942016
- [Background] Kiesel K, Plisky P, Butler R. Functional movement test scores improve following a standardized off-season intervention program in professional football players. Scand J Med Sci Sports. 2011 Apr;21(2):287-92. doi: 10.1111/j.1600-0838.2009.01038.x. PMID 20030782
- [Background] Caraffa A, Cerulli G, Projetti M, Aisa G, Rizzo A. Prevention of anterior cruciate ligament injuries in soccer. A prospective controlled study of proprioceptive training. Knee Surg Sports Traumatol Arthrosc. 1996;4(1):19-21. doi: 10.1007/BF01565992. PMID 8963746
- [Background] McGuine TA, Keene JS. The effect of a balance training program on the risk of ankle sprains in high school athletes. Am J Sports Med. 2006 Jul;34(7):1103-11. doi: 10.1177/0363546505284191. Epub 2006 Feb 13. PMID 16476915
- [Background] Lisman P, Nadelen M, Hildebrand E, Leppert K, de la Motte S. Functional movement screen and Y-Balance test scores across levels of American football players. Biol Sport. 2018 Sep;35(3):253-260. doi: 10.5114/biolsport.2018.77825. Epub 2018 Aug 27. PMID 30449943
- [Background] Wong TKK, Ma AWW, Liu KPY, Chung LMY, Bae YH, Fong SSM, Ganesan B, Wang HK. Balance control, agility, eye-hand coordination, and sport performance of amateur badminton players: A cross-sectional study. Medicine (Baltimore). 2019 Jan;98(2):e14134. doi: 10.1097/MD.0000000000014134. PMID 30633230
- [Background] Sipe CL, Ramey KD, Plisky PP, Taylor JD. Y-Balance Test: A Valid and Reliable Assessment in Older Adults. J Aging Phys Act. 2019 Sep 1;27(5):663-669. doi: 10.1123/japa.2018-0330. PMID 30676192